CLINICAL TRIAL: NCT06230757
Title: Effects of Psilocybin With Psychological Support on Anhedonia in Treatment-resistant Depression: a Randomized Controlled Pilot Trial
Brief Title: Psilocybin for Treatment-Resistant Depression
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22-1681
Record Dates: First submitted 2024-01-19; First posted 2024-01-30 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Major Depressive Disorder; Anhedonia; Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Major; Anhedonia; Depressive Disorder, Treatment-Resistant | interventions — Psilocybin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Psilocybin (Experimental): Participants receive Psilocybin 25mg capsule orally, administered with psychological support, on dosing day.
  Interventions: Drug: Psilocybin 25mg
- Active Placebo (Placebo Comparator): Participants receive Psilocybin 1mg capsule (identical to the Psilocybin 25mg capsule) orally, administered with psychological support, on dosing day.
  Interventions: Drug: Placebo (active placebo)

INTERVENTIONS:
Drug: Psilocybin 25mg — 25mg psilocybin capsule
  Arms: Psilocybin
Drug: Placebo (active placebo) — 1mg psilocybin capsule
  Other Names: Ultra Low Dose Psilocybin
  Arms: Active Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of psilocybin on the symptom of anhedonia in individuals with treatment-resistant major depressive disorder.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 21 years of age at Screening
* Diagnosis of Major Depressive Disorder (MDD)
* Score of at least 12 (symptomatic depression) on administration of the Montgomery Asberg Depression Rating Scale (MADRS)
* Score of at least a 3 on question 8 on the MADRS evaluating loss of interest and ability to feel at both Screening and Baseline Visit 1
* The participant's Major depressive disorder meets the criteria for being treatment-resistant, defined as not experiencing a 50% improvement to two or more antidepressant treatments for adequate duration (6 weeks minimum) within the current episode, as determined by the Antidepressant Treatment Response Questionnaire (Desseilles et al., 2011; Posternak et al., 2004)
* Sufficiently competent in English Language
* Currently under the care of a psychiatric practitioner (MD, DO, NP, PA) OR under the consistent care of a clinician within the UCHealth/CUMedicine health system (for example, primary care provider, neurologist, therapist). Participants engaged in additional psychosocial treatments beyond seeing a psychiatric practitioner or regular therapist will be evaluated on a case by case basis.
* Right-handed
* Women of childbearing potential (WOCBP) must agree to practice an effective means of birth control throughout the duration of the study. A person of childbearing potential is anyone born female who has experienced menarche and who has not undergone surgical sterilization (eg, hysterectomy, bilateral salpingectomy, bilateral oophorectomy) or has not completed menopause. Menopause is defined clinically as 12 months of amenorrhea in a person over age 45 in the absence of other biological, physiological, or pharmacological causes.
* Have an identified support person and agree to be accompanied home (or to an otherwise safe destination) by the support person, or another responsible party, following dosing
* Written informed consent obtained from participant and ability for subject to comply with the requirements of the study.
* Ability to abstain from caffeine and nicotine for 2 hours prior to fMRI scan visits

Exclusion Criteria:

* Unstable medical conditions or serious abnormalities of complete blood count, chemistries, or EKG that in the opinion of the study physician would preclude safe participation in the trial. Some examples include:

  1. Congestive heart failure
  2. Clinically significant arrhythmias (e.g. ventricular fibrillation, torsades) or clinically significant EKG abnormality (i.e. QTC interval > 450)
  3. Recent acute myocardial infarction or evidence of ischemia
  4. Malignant hypertension
  5. Congenital long QT syndrome
  6. Acute renal failure
  7. Severe hepatic impairment
  8. Respiratory failure
* Risk for hypertensive crisis defined as Screening, Baseline, and Medication Session (prior to dosing) Blood Pressure >140/90 mmHg.
* High resting heart rate defined as Screening, Baseline, and Medication Session (prior to dosing) heart of rate of >90 BPM
* Significant CNS pathology as determined by self-report and confirmed by a history and physical examination and review of medical records. Current and historical psychiatric disorders will be determined by the MINI. Specific examples include:

  1. Primary or secondary cerebral neoplasm
  2. Epilepsy
  3. History of stroke
  4. Cerebral aneurysm
  5. Dementia
  6. Delirium

  h. Current or lifetime primary psychotic disorder, bipolar affective disorder, affective disorder with psychotic features. Some examples include: i. Schizophrenia spectrum disorders j. Schizoaffective disorder k. Bipolar I or Bipolar II disorder l. History of mania m. Major depressive disorder with psychotic features
* Family history of first-degree relative with psychotic or serious bipolar spectrum illnesses. Examples include first-degree relative with:

  1. Schizophrenia spectrum disorders
  2. Schizoaffective disorder
  3. Bipolar I disorder with psychotic features
* High risk of adverse emotional or behavioral reaction based on investigator's clinical evaluation. Examples include:

  1. Agitation
  2. Violent behavior
* Active SUDs evaluated by the MINI and defined as: DSM-5 criteria for moderate or severe alcohol or drug use disorder (excluding caffeine and nicotine) within the past year
* Extensive use of serotonergic hallucinogens (e.g. LSD, psilocybin) defined as:

  1. Any use in the last 6 months
  2. >25 lifetime uses
* History of hallucinogen persisting perception disorder (HPPD)
* Women who are pregnant, as indicated by a positive urine pregnancy test at Screening. Women who intend to become pregnant during the study or who are currently nursing.
* History of severe suicide attempt requiring hospitalization in the past year
* Have any suicidal ideation or thoughts, in the opinion of the study physician or PI, that presents a serious risk of imminent suicidal or self-injurious behavior
* Use of drugs or dietary supplements that per the discretion of the study team, have a mechanism of action that would interfere with procedures of study or have an adverse interaction with the study drug. Examples include direct agonists/antagonists of serotonin receptors such as those listed below. Selective Serotonin Re-uptake Inhibitors and Serotonin Norepinephrine Re-uptake Inhibitors are allowed at the discretion of the PI. Individuals need to be off all non-allowed drugs for a period of 5 half-lives prior to the baseline visit.

  1. Antipsychotics
  2. Trazodone
  3. Nefazodone
  4. Cyproheptadine
  5. Mirtazapine
  6. Flibanserin
  7. Tricyclic antidepressants
  8. Monoamine oxidase inhibitors
  9. Lithium
  10. Efavirenz
  11. Serotonergic dietary supplements including St. John's Wort, L-tryptophan and 5-Hydroxytryptophan (5-HTP)
* Psychiatric condition judged to be incompatible with establishment of rapport with therapy team and/or safe exposure to psilocybin based on investigator's clinical evaluation
* Have an allergy or intolerance to any of the materials contained in either drug product
* Have a positive urine drug test including Amphetamines, Barbiturates, Buprenorphine, Benzodiazepines, Cocaine, Methamphetamine, MDMA, Methadone, Opiates (Morphine, Oxycodone), Phencyclidine (PCP).

  1. Note: Prescribed benzodiazepine medications and non-benzodiazepine sleeping medications will be allowed to continue through the study period for participants who have been on a stable dose of such a medicine for at least 6 weeks prior to Screening, as determined during review of concomitant medications.
  2. Note: Participants using cannabis, including legal cannabis, for any purposes and who do not screen positive for a moderate to severe substance use disorder must agree to refrain from use beginning at Screening and through to the end of the study.
  3. Note: Participants using prescribed psychostimulants (amphetamines and Ritalin), must agree to refrain from use for five half-lives of the drug as confirmed with a negative Baseline drug test, and through to the end of the study.
* Have any psychological or physical symptom, medication or other relevant finding prior to baseline visit based on the clinical judgment of the PI or relevant clinical study staff that would make a participant unsuitable for the study.
* Claustrophobia
* Lack of internet access
* Weight over 300 pounds
* Metal in body unsafe for MRI or conditions that would make MRI unsafe for participants (e.g. aneurysm clip, cardiac pacemaker, etc.).
* Known contraindication to the drugs clonidine, diazepam, or olanzapine including:

  1. Hypersensitivity or allergy to clonidine, diazepam, or olanzapine
  2. Myasthenia gravis
  3. Severe respiratory insufficiency
  4. Severe hepatic insufficiency
  5. Acute narrow-angle glaucoma 23. History of valvular heart disease 24. Inability of the study team to obtain proper medical/psychiatric information (e.g. records from a current or previous clinician), that per the PI, would prevent an adequate assessment of the patient's eligibility and ability to safely participate in the study.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-08 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in self-reported anhedonia scores on the Dimensional Anhedonia Rating Scale (DARS). | One week post-dosing
  The DARS is a 17-item scale that captures multiple domains of anhedonia found in depression. Scores range from 0 to 68 with lower scores indicating greater anhedonia and 68 indicating no anhedonia.

SECONDARY OUTCOMES:
Change from baseline in self-reported anhedonia scores on the Dimensional Anhedonia Rating Scale (DARS). | Eight weeks post-dosing
  The DARS is a 17-item scale that captures multiple domains of anhedonia found in depression. Scores range from 0 to 68 with lower scores indicating greater anhedonia and 68 indicating no anhedonia.
Change from baseline in self-reported anhedonia scores on the Snaith-Hamilton Pleasure Scale (SHAPS). | One week and eight weeks post-dosing
  The SHAPS is a 14-item scale that assesses the pleasure component of hedonic experience across multiple domains. Scores range from 0 to 14 with 0 indicating no anhedonia and high scores indicating greater anhedonia.
Change from baseline in response bias for the high reward condition on the Probabilistic Reward Task (PRT) | One and eight weeks post-dosing
  The PRT is a behavioral task that assesses the capacity to develop a response bias towards more highly rewarded stimuli, in which individuals with MDD demonstrate reduced bias towards highly rewarded stimuli.
Change from baseline in nucleus accumbens neural activation during expectation of reward versus expectation of non-reward during the Monetary Incentive Delay Task (MID). | One week post-dosing
  The MID is used in conjunction with fMRI to assess neural activity during reward processing and reliably induces neural activation in brain regions related to reward.
Change from baseline in depression scores of the clinician-rated Montgomery-Asberg Depression Rating Scale (MADRS). | One and eight weeks post-dosing
  The MADRS is a standard 10-item clinician-rated scale that assesses severity of depression in anti-depressant trials. Scores range form 0-60, with scores of 0-6 indicating no depression, 7-19 indicating mild depression, 20-34 indicating moderate depression and 35 or greater indicating severe depression.
Change from baseline in depression scores as measured by self-report on the Quick Inventory of Depressive Symptomatology (QIDS-SR-16). | One, four, and eight weeks post-dosing
  The QIDS-SR-16 is a widely used 16-item self-report scale of depressive symptoms. Scores range form 0-27, with scores of 0-5 indicating no depression, 6-10 indicating mild depression, 11-15 indicating moderate depression, 16-20 indicating severe depression, and 21-27 indicating very severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Novick, MD, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No